CLINICAL TRIAL: NCT04046042
Title: Virtual Reality Exercise Intradialysis: Tolerance and Dialysis Dose Effects During the Last vs. First Part of the Hemodialysis Session
Brief Title: Virtual Reality Intradialysis: Last vs. First Part of the Session
Acronym: VRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de Manises (Other); Universitat Politècnica de Valéncia (Unknown)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReVID
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease on Dialysis; Hemodialysis Complication
Keywords: Exercise; Virtual reality; physical function; health-related quality of life; hemodynamic instability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two exercise groups, during the first two hours of hemodialysis or during the last two hours of hemodialysis
Who Masked: Investigator, Outcomes Assessor
Masking Description: A team of assessors, different from the researchers implementing the exercise, will record all dependent variables. A blind researcher will randomize participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise time (Active Comparator): During 12 months subjects will exercise during the first two hours of the hemodialysis session. A virtual reality exercise program will be implemented
  Interventions: Other: Conventional exercise
- Experimental group (Experimental): During 12 months subjects will exercise during the last two hours of the hemodialysis session. A virtual reality exercise program will be implemented
  Interventions: Other: Exercise during the last two hours of the hemodialysis session

INTERVENTIONS:
Other: Conventional exercise — Virtual reality exercise performed during the first two hours of the hemodialysis session
  Arms: Conventional exercise time
Other: Exercise during the last two hours of the hemodialysis session — Virtual reality exercise performed during the last two hours of the hemodialysis session
  Arms: Experimental group

SUMMARY:
The main objective of this investigation is to assess if an intradialysis virtual reality exercise program during the last two hours of the hemodialysis session results in greater hemodynamic stability than exercise performed during the first two hours of the hemodialysis session.

The secondary aims are to assess the impact of intradialysis virtual reality exercise during the last two hours of the hemodialysis session on dialysis efficacy, postdialysis molecules rebound, adherence to exercise, functional capacity, physical activity level, health-related quality of life, cognitive function, morbidity, frailty and dependency. We will also analyze the reliability of muscle strength assessment of lower limb muscles with a handheld dynamometer during hemodialysis.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups. The first group will perform a virtual reality exercise during the first two hours of the hemodialysis session. The second group will perform a virtual reality exercise during the last two hours of the hemodialysis session. The exercise program will last for 9 months.

The virtual reality exercise will undertake up to 30 minutes of exercise. After warming up, participants will play to an adapted 'treasure hunt' game. Their legs movements will be the players projected into an individual tv that will give them feedback regarding their achievements. The aim of the game will be to achieve the higher possible score. They will move their legs to pick up coins and to avoid bombs. An adapted Kinect technology will be used for game development. The exercise session will end-up with a cool-down period that will include simple lower limb stretching exercises. Two more games will be introduced progressively for patients not to get bored, 'Air Hockey' and 'Simon'.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months in hemodialysis treatment
* Clinically stable

Exclusion Criteria:

* Recent cardiac events (less than 3 months)
* Unable to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-08-29 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of hypotension episodes | 3 Months
  Number of hypotension episodes, including hypotension that requires treatment, hypertensive crisis and acute arrhythmias
Number of hypotension episodes | 6 Months
  Number of hypotension episodes, including hypotension that requires treatment, hypertensive crisis and acute arrhythmias
Number of hypotension episodes | 12 Months
  Number of hypotension episodes, including hypotension that requires treatment, hypertensive crisis and acute arrhythmias

SECONDARY OUTCOMES:
Change from baseline postdialysis rebound urea, creatinine, phosphorus and potassium at 3 months | Baseline and 3 months
  Postdialysis rebound urea, creatinine, phosphorus and potassium. All measurements presented as a percentage.
Change from baseline dialysis dose at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Dialysis dose, measured through Kt/V
Adherence, as number of sessions performed /number of sessions offered | Baseline, 3 Months, 6 months and 12 months
  Sessions performed/sessions offered
Change from baseline short physical performance battery at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Score achieved at the battery that includes balance tests (4 points), sit to stand to sit 5 (4 points) and and gait speed (4 points). The total score is calculated , from 1 to 12, being 12 the highest functional score
Change from baseline gait speed at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Speed to cover 4 meters, in meters/second
Change from baseline handgrip at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Bilateral handgrip strength
Change from baseline lower limb muscle strength at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Muscle strength measured with a handheld dynamometer on the main muscle groups during hemodialysis
Change from baseline one-leg standing test at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Time achieved while standing on one leg
Change from baseline sit to stand 10 test at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Time to perform 10 repetitions sit to stand
Change from baseline sit to stand 60 at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Sit to stand repetitions performed in 60 seconds
Change from baseline timed up and go at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Time to stand up, walk 3 meters, come back and sit down again
Change from baseline one-leg heel rise test at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Number of heel rise repetitions achieved
Change from baseline 6 minutes walk test at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Number of meters walked in 6 minutes
Change from baseline Physical activity level at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Physical activity questionnaires
Change from baseline Health related quality of life at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Medical outcomes survey Short Form 36 questionnaire to measure health-related quality of life, rated from 0 to 100, being the highest score the better the quality of life
Change from baseline Cognitive function at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Mini-mental State Examination questionnaire, score ranges from 0 to 30, higher scores indicates higher cognitive function
Change from baseline disability by Barthel Index at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Functional evaluation by Barthel Index, to evaluate capacity to perform daily tasks without assistance. Score ranges from 0 to 100. Higher scores indicates higher capacity to perform activities.
Change from baseline frailty (slowness; weakness; weight loss/malnutrition;low physical activity; exhaustion) at 3 months, 6 months, and 12 months | Baseline, 3 Months, 6 months and 12 months
  Frailty will be measured from 0 to 5, depending on how many of the 5 components are present in each subject, being 5 the highest frailty score

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura-Ortí, PhD, Principal Investigator — Universidad CEU Cardenal Herrera, UCH CEU
Locations (1):
- Hospital de Manises, Manises, Valencia, Spain

REFERENCES:
- [Background] Segura-Orti E, Perez-Dominguez B, Ortega-Perez de Villar L, Melendez-Oliva E, Martinez-Gramage J, Garcia-Maset R, Gil-Gomez JA. Virtual reality exercise intradialysis to improve physical function: A feasibility randomized trial. Scand J Med Sci Sports. 2019 Jan;29(1):89-94. doi: 10.1111/sms.13304. Epub 2018 Oct 7. PMID 30230041
- [Background] Segura-Orti E, Garcia-Testal A. Intradialytic virtual reality exercise: Increasing physical activity through technology. Semin Dial. 2019 Jul;32(4):331-335. doi: 10.1111/sdi.12788. Epub 2019 Mar 27. PMID 30916415
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Background] Segura-Orti E, Johansen KL. Exercise in end-stage renal disease. Semin Dial. 2010 Jul-Aug;23(4):422-30. doi: 10.1111/j.1525-139X.2010.00766.x. PMID 20701722
- [Background] Segura-Orti E. [Exercise in haemodyalisis patients: a literature systematic review]. Nefrologia. 2010;30(2):236-46. doi: 10.3265/Nefrologia.pre2010.Jan.10229. Epub 2010 Jan 21. Spanish. PMID 20098466
- [Background] Garcia Testal A, Garcia Maset R, Hervas Marin D, Perez-Dominguez B, Royo Maicas P, Rico Salvador IS, Melendez-Oliva E, Molina Aracil J, Murgui Chiva M, Del Pozo Blanco O, Olague Diaz P, Fernandez Najera JE, Torregrosa De Juan E, Benedito Carrera C, Segura-Orti E. Influence of Physical Exercise on the Dialytic Adequacy Parameters of Patients on Hemodialysis. Ther Apher Dial. 2019 Apr;23(2):160-166. doi: 10.1111/1744-9987.12762. Epub 2018 Oct 19. PMID 30226299
- [Background] Ortega-Perez de Villar L, Martinez-Olmos FJ, Junque-Jimenez A, Amer-Cuenca JJ, Martinez-Gramage J, Mercer T, Segura-Orti E. Test-retest reliability and minimal detectable change scores for the short physical performance battery, one-legged standing test and timed up and go test in patients undergoing hemodialysis. PLoS One. 2018 Aug 22;13(8):e0201035. doi: 10.1371/journal.pone.0201035. eCollection 2018. PMID 30133445
- [Background] Segura-Orti E, Kouidi E, Lison JF. Effect of resistance exercise during hemodialysis on physical function and quality of life: randomized controlled trial. Clin Nephrol. 2009 May;71(5):527-37. doi: 10.5414/cnp71527. PMID 19473613
- [Background] Segura-Orti E, Rodilla-Alama V, Lison JF. [Physiotherapy during hemodialysis: results of a progressive resistance-training programme]. Nefrologia. 2008;28(1):67-72. Spanish. PMID 18336134